CLINICAL TRIAL: NCT06662968
Title: A Study on Early Sucking of Lollipops in Preschool Children After Adenotonsillectomy:a Randomized Controlled Trial
Brief Title: A Study on Early Sucking of Lollipops in Preschool Children After Adenotonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maternal and Child Health Hospital of Hubei Province (Other)
Responsible Party: Principal Investigator, Li Na, Deputy Chief Physician, Maternal and Child Health Hospital of Hubei Province
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCHH_006
Record Dates: First submitted 2024-10-21; First posted 2024-10-29 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Adenotonsillectomy
Keywords: Lollipops; Adenotonsillectomy
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lollipop group (Experimental): Lollipop group patients were given lollipops for sucking in the PACU
- Control group (Active Comparator): Control group patients were received routine nursing treatment in the PACU.

INTERVENTIONS:
Other: Lollipop group — In the Lollipop group,children were sent to the recovery room (PACU) for observation after extubation after surgery.They were given lollipops for sucking without chewing after waking up.Throughout the entire sucking process, we continuously monitor vital signs.
Other: Control group — In the Control group,children were sent to the recovery room (PACU) for observation after extubation after surgery.They were received routine nursing treatment.

SUMMARY:
The aim of this study is to observe the consumption effect of early lollipop sucking in preschool children after adenotonsillectomy through clinical experiments, and to explore the impact of early postoperative lollipop consumption on postoperative agitation, incidence of postoperative nausea and vomiting, and postoperative wound recovery rate.

Participants will be randomly allocated to two groups:a lollipop sucking group (Group A) and a control group (Group B), Two groups of children were sent to the recovery room (PACU) for observation after extubation . Group A patients were given lollipops for sucking after waking up, while Group B received routine nursing treatment.

The goal of this clinical trial is to explore whether lollipops have advantages in early postoperative feeding and alleviating postoperative agitation in children, and to provide reliable clinical evidence for the consumption of lollipops after surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who choose to have adenotonsillectomy surgery
* the American Society of Anesthesiologists (ASA) physical status ranked I-II
* competent to provide informed consent

Exclusion Criteria:

* psychiatric disorders
* upper respiratory tract infection
* high risk of reflux aspiration
* carbohydrate malabsorption syndrome and other endocrine or genetic metabolic diseases (contraindications of lollipop ingredients)

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-04-28 (Actual); Study Completion 2025-04-28 (Actual)

PRIMARY OUTCOMES:
Postoperative agitation score | Time Frame: intraoperative period,10 minutes-1 hours
  Postoperative agitation score will be recorded at 6 time points, including the time of entering the recovery room (Time 0), when the lollipop is given (Time 1), when the lollipop is given for 10 minutes(Time 2), when the lollipop is given for 20 minutes(Time 3), when the lollipop is given for 30 minutes(Time 4) and leave the recovery room (T5).
Incidence of nausea and vomiting | Postoperative 1 minute-5hours
  Incidence of nausea and vomiting will be recorded during the time of the recovery room and four hours after returning to the ward .

SECONDARY OUTCOMES:
Spo2 | Postoperative 1 minute - 5hours
  Spo2 will be continuous monitoring and recorded during the time of the recovery room
other adverse reactions | Postoperative 10 minutes - 3days
  The occurrence of adverse reactions( wound infection and others) were continuous monitoring and recorded after the operation
the time of leaving the recovery room and the hospital | Postoperative 1 hour - 3days
  the time of leaving the recovery room and the hospital will be recorded
family satisfaction | Postoperative 5 hours
  Record the satisfaction of the parents with this operation ,defined as a score out of 100

CONTACTS AND LOCATIONS:
Overall Officials: Na Li, MD, Principal Investigator — Maternal and Child Health Hospital of Hubei Province
Locations (1):
- Maternal and Child Health Hospital of Hubei Province, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes